CLINICAL TRIAL: NCT01116895
Title: An International, Multi-centre, Prospective, Randomised, Double-blind, 4-arm, Placebo Controlled, Parallel Group Study With 12 Weeks Once Daily Oral Treatment in Subjects With Psoriasis Vulgaris
Brief Title: A Proof of Concept Study Comparing Three Doses of an Oral Solution of LEO 22811 With a Placebo Oral Solution for the Treatment of Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 22811-S22
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis Vulgaris; Systemic; Anti-psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LEO 22811 0.5 mg (Active Comparator): LEO 22811 0.5 mg: Oral solution
  Interventions: Drug: LEO 22811
- LEO 22811 1.5 mg (Active Comparator): LEO 22811 1.5 mg: Oral solution
  Interventions: Drug: LEO 22811
- LEO 22811 3.0 mg (Active Comparator): LEO 22811 3.0 mg: Oral solution
  Interventions: Drug: LEO 22811
- Placebo (Placebo Comparator): Placebo: Oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 22811 — Oral solution
  Arms: LEO 22811 0.5 mg; LEO 22811 1.5 mg; LEO 22811 3.0 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
An international, multi-centre, prospective, randomised, double-blind, 4-arm, placebo controlled, parallel group study with 12 weeks once daily oral treatment in subjects with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Following verbal and written information about the trial the subject must provide signed and dated informed consent before any study related activity is carried out, including activities relating to the washout period.
* Clinical diagnosis of psoriasis vulgaris, for at least 6 months prior to randomisation, and currently covering at least 10% of the body surface area (BSA)
* Candidates for systemic anti-psoriatic treatment
* Psoriasis Area and Severity Index (PASI) ≥10
* Disease severity of moderate, severe or very severe according to the Investigators' Global Assessment of disease severity (IGA)
* Aged 18 years or above
* Any race or ethnicity
* Males, surgically sterile females (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or post menopausal females (at least 1 year since last menses)
* Attending hospital outpatient clinic or the private practice of a dermatologist

Exclusion Criteria:

* Systemic treatment with biological therapies whether marketed or not with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * Etanercept - 4 weeks
  * Adalimumab, alefacept, infliximab - 2 months
  * Ustekinumab - 4 months
* Systemic treatment with all other therapies (other than biologics) with a possible effect on psoriasis vulgaris (e.g.corticosteroids, retinoids, immunosuppressants, methotrexate, cyclosporin or fumaric acid) within 4 weeks prior to randomisation
* PUVA therapy within 4 weeks prior to randomisation
* UVB therapy within 2 weeks prior to randomisation
* Any topical treatment (except for emollients/ medicated shampoo) within 2 weeks prior to randomisation
* Initiation of, or changes to concomitant medication that could affect psoriasis vulgaris (e.g. beta-blockers, anti-malaria drugs, lithium) 2 weeks prior to randomisation and during the study
* Current diagnosis with erythrodermic, exfoliative or pustular psoriasis
* Other current skin conditions that may confound the evaluation of psoriasis vulgaris as judged by the Investigator
* Generally in good health and does not have any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, haematologic, or gastrointestinal disease, immunologic insufficiency, or other major diseases or current condition which, in the opinion of the Investigator, would put the subject at risk by participating in the study
* Current active tuberculosis or latent tuberculosis
* Planned exposure to the sun during the study that may affect psoriasis vulgaris
* Known malignancy or history of malignancy (other than cervical carcinoma in situ, basal cell or squamous cell carcinoma) within the 5 year period prior to randomisation
* Live vaccination within the 4 weeks prior to randomisation
* Males who do not agree to use adequate contraception during the study (including follow-up) to ensure their partner does not become pregnant
* Known or suspected hypersensitivity to component(s) of the investigational product
* Current participation in any other interventional trial
* Treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within 4 weeks or 5 half-lives (whichever is longer) prior to randomisation
* Previously randomised in this study
* Known or, in the opinion of the Investigator, is unlikely to comply with the Clinical Study Protocol (e.g., alcohol abuse, drug dependency or psychotic state).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Poulin, MD, Principal Investigator — Centre de Recherche Dermatologique du Quebec Metropolitain
Locations (2):
- Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Canada
- Hôpital Saint-Louis, Service de Dermatologie, Paris, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg | Placebo
Started | 16 | 15 | 18 | 14
Completed | 12 | 8 | 14 | 11
Not Completed | 4 | 7 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 18 | 14 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (9.3) | 49.8 (14.1) | 42.4 (13.6) | 44.9 (12.0) | 46.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 1 | 11
  Male | 14 | 11 | 14 | 13 | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7 | 8 | 8 | 7 | 30
  France | 9 | 7 | 10 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Psoriasis Area and Severity Index (PASI)
Description: The investigator made assessments of the extent and severity of clinical signs of the participant's psoriasis on specific areas of the body in terms of three clinical signs: redness, thickness and scaliness.
  The extent of psoriatic involvement was recorded for each of four areas; head, arms, trunk and legs using the following scale:
  0. = no involvement
  1. = <10%
  2. = 10-29%
  3. = 30-49%
  4. = 50-69%
  5. = 70-89%
  6. = 90-100%
  For each clinical sign a single score (0, 1, 2, 3 or 4) reflecting the average severity of all psoriatic lesions on the given body region was determined.
  PASI was calculated based on the investigator's assessment of the disease locally (head, trunk, arm, legs) using the following formula:
  Head: 0.1 (R + T + S)E = W Arms: 0.2 (R + T + S)E = X Trunk: 0.3 (R + T + S)E = Y Legs: 0.4 (R + T + S)E = Z R = score for redness; T = score for thickness, S = score for scaliness; E = score for extent The sum of W+X+Y+Z gives the total PASI that ranges from 0 to 72.
Time Frame: Baseline (Day 0) to end of treatment (Day 84)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of change in PASI index score
Arm/Group | Placebo | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg
Number analyzed (Participants) | 14 | 16 | 15 | 18
percentage of change in PASI index score | -5.6 (44.9) | -7.6 (29.1) | -0.3 (43.5) | -12.7 (45.2)
Statistical Analysis 1: Comparison: Placebo vs LEO 22811 0.5 mg; Test type: Other; p = 0.89, ANOVA; Least square mean difference = -2.2, 95% CI 2-sided [-32.6 to 28.2]
Statistical Analysis 2: Comparison: Placebo vs LEO 22811 1.5 mg; Test type: Other; p = 0.77, ANOVA; Least square mean difference = 4.5, 95% CI 2-sided [-26.2 to 35.3]
Statistical Analysis 3: Comparison: Placebo vs LEO 22811 3.0 mg; Test type: Other; p = 0.65, ANOVA; Least square mean difference = -6.7, 95% CI 2-sided [-36.2 to 22.8]

2. Secondary Outcome: Participants With at Least 75% Reduction in PASI (PASI 75)
Time Frame: From baseline (Day 0) to end of treatment (Day 84)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg
Number analyzed (Participants) | 14 | 16 | 15 | 18
Participants
  Yes | 0 | 1 | 0 | 2
  No | 14 | 15 | 15 | 16

3. Secondary Outcome: Participants With at Least 50% Reduction in PASI (PASI 50)
Time Frame: From baseline (Day 0) to end of treatment (Day 84)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg
Number analyzed (Participants) | 14 | 16 | 15 | 18
Participants
  Yes | 2 | 1 | 2 | 4
  No | 12 | 15 | 13 | 14

4. Secondary Outcome: Participants With "Controlled Disease" According to the Investigators' Global Assessment (IGA)
Description: At Visits 1 to 8 the investigator made a global assessment of the disease severity (IGA) using a 6-point scale (clear, almost clear, mild, moderate, severe, very severe). This assessment represents average lesion severity on head, trunk, arm and legs. The assessment was based on the condition of the disease at the time of evaluation and not in relation to the condition at a previous visit. Participants classified as clear or almost clear according to IGA was considered to have "controlled disease".
Time Frame: At end of treatment (Day 84)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg
Number analyzed (Participants) | 14 | 16 | 15 | 18
Participants
  Controlled | 0 | 0 | 0 | 1
  Non-controlled | 14 | 16 | 15 | 17

5. Secondary Outcome: Participants With Satisfactory Response According to IGA
Description: "Satisfactory response" was defined as participants classified as "Clear" or "Almost Clear" or "Mild" according to the IGA.
Time Frame: At end of treatment (Day 84)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg
Number analyzed (Participants) | 14 | 16 | 15 | 18
Participants
  Satisfactory | 2 | 1 | 1 | 2
  Unsatisfactory | 12 | 15 | 14 | 16

ADVERSE EVENTS:
Time Frame: From Day 0 to Follow-up (Day 122 + 28±2 days)
Arm/Group | Placebo | LEO 22811 0.5 mg | LEO 22811 1.5 mg | LEO 22811 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16 | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/16 | 1/15 | 0/18
Other Adverse Events (participants affected / at risk) | 10/14 | 11/16 | 11/15 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | LEO 22811 0.5 mg (N=16) | LEO 22811 1.5 mg (N=15) | LEO 22811 3.0 mg (N=18)
Proteinurea (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | LEO 22811 0.5 mg (N=16) | LEO 22811 1.5 mg (N=15) | LEO 22811 3.0 mg (N=18)
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 0 | 1
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 2
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Bacillary angiomatosis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 1 | 1 | 0 | 1
Gastrointestinal fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3 | 2
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vaginal mycosis (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 1 | 0 | 1
C-reactive protein increased (Investigations) | 2 | 3 | 0 | 2
Electrocardiogram normal (Investigations) | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 1 | 1
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0
Mean cell volume increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 1
Platelet count increased (Investigations) | 1 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Ganglion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 4
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0
Stress symptoms (Psychiatric disorders) | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual publications or presentations of data by one or more Investigator(s) shall not be made before the results of the joint publication have been made public. The company retains the right to have any publication submitted to the company for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.